CLINICAL TRIAL: NCT05939583
Title: Effect of Shock Wave Therapy on Upper Trapezius Trigger Points in Patients With Cervicogenic Headache. a Randomized Controlled Trial
Brief Title: Effect of Shock Wave Therapy on Upper Trapezius Trigger Points in Patients With Cervicogenic Headache.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Ahmed Magdy Alshimy, Lecturer Of Neurological Physical Therapy - Faculty Of Physical Therapy - October 6 University, October 6 University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: REC/2111/MTI.PT/2303123
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Cervicogenic Headache
Keywords: Shock wave therapy; Trapezius trigger points; Cervicogenic headache
MeSH Terms: conditions — Post-Traumatic Headache | interventions — Extracorporeal Shockwave Therapy; Transcutaneous Electric Nerve Stimulation; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): The treatment group will receive US, TENS, IR and exercises in addition to shock waves therapy. Patients will receive 3 sessions per week for 4 weeks
  Interventions: Other: Shock Wave Therapy; Other: US, TENS, IR and exercises.
- Control Group (Experimental): Control group will receive US, TENS, IR and exercises. Patients will receive 3 sessions per week for 4 weeks
  Interventions: Other: US, TENS, IR and exercises.

INTERVENTIONS:
Other: Shock Wave Therapy — Receiving Shock wave therapy + US, TENS, IR and exercises.
  Other Names: US, TENS, IR and exercises.
  Arms: Treatment Group
Other: US, TENS, IR and exercises. — Receiving US, TENS, IR and exercises only.

SUMMARY:
Control group will receive US, TENS, IR and exercises. The treatment group will receive the same program in addition to shock waves therapy. Patients will receive 3 sessions per week for 4 weeks.

DETAILED DESCRIPTION:
Control group will receive US, TENS, IR and exercises. The treatment group will receive the same program in addition to shock waves therapy. Patients will receive 3 sessions per week for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Fifty patients from both genders.
* Age ranging from 20 to 40 years.
* Referred by an orthopedist with a diagnosis of Mechanical neck dysfunction (MND) to physical therapy at the outpatient clinic of the Faculty of Physical Therapy, MTI University.

Exclusion Criteria:

* All other disorders.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | 4 weeks
  Assess degree of pain from 1 (No Pain) to 10 (Severe Pain)
Neck disability index | 4 weeks
  Assess degree of neck disability.
Kinesiological EMG | 4 weeks
  Analysis of root mean square for upper trapezius muscle functions.
Kinesiological EMG | 4 weeks
  Analysis of median frequency for upper trapezius muscle functions.

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University, El-Sheikh Zayed City, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No